CLINICAL TRIAL: NCT00200525
Title: A Randomized, Placebo-Controlled Study of the Continued Efficacy and Safety of SC Apomorphine in the Treatment of Off Episodes in Patients With "On/Off" or "Wearing-Off" Effects Associated With Late-Stage PD After Apomorphine Use
Brief Title: Continued Efficacy and Safety of Apomorphine in Patients With Late-Stage Parkinsons Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APO302
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

INTERVENTIONS:
Drug: apomorphine HCl injection

SUMMARY:
Study to measure the continued effectiveness of apomorphine after previous exposure of at least three months duration.

ELIGIBILITY:
Inclusion Criteria:

* Adults of any age ≥ 18
* Men and non-pregnant, non-lactating women
* Women of childbearing potential had a negative serum (Beta HCG) pre-study pregnancy test prior to randomization
* Women of childbearing potential used an acceptable form of contraception
* Patients with a clinical diagnosis of idiopathic Parkinson's Disease, i.e., not induced by drugs or caused by other diseases;
* Patients classified as stage (II-IV) of the Hoehn and Yahr scale for staging the severity of Parkinson's Disease
* The patient must have been on an optimally maximized oral therapy regimen. Optimized oral anti-parkinson medications must have included levodopa/carbidopa inhibitors, in either immediate or delayed release forms, plus at least one direct acting oral dopamine agonist for at least 30 days prior to randomization
* Patients must have been receiving apomorphine subcutaneous injections for rescue therapy for Off events for at least three months
* The minimum apomorphine baseline-dosing requirement was an average of at least 2 doses per day over the week prior to enrollment.
* Patients participating in protocol APO401, an open-label study primarily designed to collect safety data, were eligible for participation in this trial without termination of participation in APO401

Exclusion Criteria:

* Patients under medical therapy for clinically significant psychoses or dementia not related to ingestion of anti-parkinson medications. (Patients with hallucinations or other central adverse reactions associated solely with anti-parkinson medications were not excluded.)
* Patients with a history of drug or alcohol dependency within one year prior to study enrollment
* Patients with unstable and clinically significant disease of cardiovascular (including orthostatic hypotension), hematologic (including Coombs' positive hemolytic anemia), hepatic, renal, metabolic, respiratory, gastrointestinal or endocrinological systems or neoplasm within the three months before the start of the study.
* Patinets with a history of true allergy to morphine or its derivatives (including apomorphine), sulfur, sulfur containing medications, sulfites, sulfates, Tigan(R)(trimethobenzamide).
* Patients treated with experimental agents (other than apomorphine intermittent subcutaneous injections) within 30 days before study entry. Patients with participation in MYLAN-sponsored study APO202 were excluded from participation in this study.
* Patients whose apomorphine regimen was characterized by administration methods other than intermittent subcutaneous injection.
* Patients who could not or would not sign an Informed Consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-07; Study Completion 2002-06

PRIMARY OUTCOMES:
Change in UPDRS Motor Score 20 minutes after dosing of apomorphine or placebo

SECONDARY OUTCOMES:
Percent change in UPDRS Motor Score from pre-dose to 10, 20, and 90 minutes after dosing
Area under the curve (AUC) for change in UPDRS Motor Score at 0, 10, 20 and 90 minutes
Time to patient-declared onset of relief (max observation time = 40 minutes)
Change in Webster Step-Seconds Test score from pre-dose to 2.5, 5, 7.5, 10, 15, 20, 40, and 90 minutes
Change in Dyskinesia Assessment from pre-dose to 10, 20 and 90 minutes after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Will Sullivan, Study Director — Mylan Bertek Pharmaceuticals